CLINICAL TRIAL: NCT00307645
Title: Mycophenolate Mofetil Versus Azathioprine for Maintenance Therapy in ANCA Associated Systemic Vasculitis
Brief Title: IMPROVE: Mycophenolate Mofetil Versus Azathioprine for Maintenance Therapy in ANCA Associated Systemic Vasculitis
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P991003
Record Dates: First submitted 2006-03-27; First posted 2006-03-28 (Estimated); Last update posted 2006-04-10 (Estimated); Status verified 2003-03

CONDITIONS: ANCA Associated Systemic Vasculitis Including Wegener's; Granulomatosis and Microscopic Polyangiitis and; Renal Limited Vasculitis
Keywords: ANCA associated systemic vasculitis; Maintenance therapy; Azathioprine; Mycophenolate mofetil
MeSH Terms: conditions — Microscopic Polyangiitis | interventions — Cyclophosphamide; Mycophenolic Acid; Azathioprine; Prednisone; Methylprednisolone

INTERVENTIONS:
Drug: Cyclophosphamide
Drug: Mycophenolate mofetil
Drug: Azathioprine
Drug: Prednisone (and methylprednisolone)

SUMMARY:
The aim of IMPROVE is to define the optimal maintenance therapy for ANCA-associated vasculitides (AASV) by comparing the AZA (standard regimen) with MMF in terms of efficacy, i.e. in preventing relapses.

HYPOTHESIS :

MMF might be more effective than azathioprine as maintenance drug in AASV patients, reducing by 50% relapse rate, with a same frequency of adverse effects

DETAILED DESCRIPTION:
AASV, including Wegener's granulomatosis (WG) and microscopic polyangiitis (MPA) and renal limited vasculitis (RLV), are progressive, multisystem, autoimmune diseases which require the prescription of immunosuppressive therapy. Treatment using corticosteroids and cytotoxic drugs has been standardised (ECSYSVASTRIAL project), but relapse rate remains high and treatment-related toxicity is non negligible. The IMPROVE trial aims to reduce this relapse rate by using mycophenolate mofetil (MMF) for maintenance therapy. The potential benefit of MMF has been suggested in a published open and uncontrolled study. Patients with newly diagnosed systemic AASV will be randomly assigned to receive either MMF or reference treatment with azathioprine (AZA), once remission has been obtained with cyclophosphamide and prednisone. MMF and AZA will be continued for a total of 42 months of therapy with concomitant prednisone dose tapering. The study will last 48 months. Hence, within the last 6 months of the study duration, the patients will not receive any immunosuppressive drugs.

The primary end-point will the disease-free period, taken as the period of time from remission until relapse or study end; secondary end-points will be adverse events, cumulative damage (assessed using damage score VDI) and immunosuppressive drug cumulative dose.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed patients with WG, MPA or renal-limited vasculitis.
* ANCA positivity. ANCA positivity requires PR3-ANCA or a typical cANCA pattern by indirect immunofluorescence (IIF), preferably confirmed by anti-PR3 ELISA. MPO-ANCA determined by ELISA requires demonstration of pANCA, and pANCA by IIF requires confirmation by anti-MPO ELISA. Optionally, central review of ANCA serology can be performed.
* Age 18 to 75 years

Exclusion Criteria:

* Any cytotoxic drug within previous year, unless started within one months of entry and according to the protocol design
* Co-existence of another systemic autoimmune disease, e.g. SLE
* Hepatitis B or Hepatitis C infection
* HIV positivity
* Failure to achieve remission after 6 months of CYC therapy
* Failure to control progressive disease with induction protocol
* Malignancy (usually exclude unless agreed with trial co-ordinator)
* Pregnancy or inadequate contraception
* Age below 18 and above 75 years*
* Endstage renal failure unless active extrarenal disease requires treatment (temporal dependency of hemodialysis is not an exclusion criterion)
* Inability for informed consent

  * After discussion with the trial administrator, patients less than 18 years may be incorporated on separate application according to the appropriate local ethic committee.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160
Dates: Start 2003-05; Study Completion 2009-08

PRIMARY OUTCOMES:
the disease-free period, defined as the time between the beginning
of the maintenance therapy (AZA or MMF) and the first relapse (minor or major)
or the end of the protocol (at 48 months)

SECONDARY OUTCOMES:
relapse rate
rate of side-effects and intolerance
cumulative doses (AZA, CS, MMF)
AUC for BVAS, SF-36 or VDI
Evolution of titers of ANCA and CRP

CONTACTS AND LOCATIONS:
Overall Officials: Loïc GUILLEVIN, MD,PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (2):
- Hopital Cochin, Paris, France
- Addenbrooke's Hospital - Departement of Medecine, Cambridge, United Kingdom

REFERENCES:
- [Derived] Morgan MD, Szeto M, Walsh M, Jayne D, Westman K, Rasmussen N, Hiemstra TF, Flossmann O, Berden A, Hoglund P, Harper L; European Vasculitis Society. Negative anti-neutrophil cytoplasm antibody at switch to maintenance therapy is associated with a reduced risk of relapse. Arthritis Res Ther. 2017 Jun 7;19(1):129. doi: 10.1186/s13075-017-1321-1. PMID 28592297
- [Derived] Hiemstra TF, Walsh M, Mahr A, Savage CO, de Groot K, Harper L, Hauser T, Neumann I, Tesar V, Wissing KM, Pagnoux C, Schmitt W, Jayne DR; European Vasculitis Study Group (EUVAS). Mycophenolate mofetil vs azathioprine for remission maintenance in antineutrophil cytoplasmic antibody-associated vasculitis: a randomized controlled trial. JAMA. 2010 Dec 1;304(21):2381-8. doi: 10.1001/jama.2010.1658. Epub 2010 Nov 8. PMID 21060104